CLINICAL TRIAL: NCT06255704
Title: A Single-arm, Single-center, Open-label Phase II Study of Zanubrutnib Combined With R-CHOP/R-DHAP Alternating Regimen for First-line MCL and Followed by Zanubrutinib Rituximab Maintenance Therapy
Brief Title: A Single-arm, Single-center, Open-label Phase II Study of Zanubrutinib Combined With R-CHOP/R-DHAP in Newly Diagnosed Mantle CellLymphoma Patients
Acronym: Z+RCHOP/RDHAP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanxi Province Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCL BTKi immunochemotherapy
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib and RCHOP/RDHAP (Experimental): Patients will receive zanubrutinib and RCHOP alternating with RDHAP for a total of 6 cycles of induction therapy, and patients who achieve complete response after 6 cycles of induction therapy will be eligible to enter a 2-year maintenance treatment period of zanubrutinib in combination with rituximab
  Interventions: Drug: Zanubrutinib and RCHOP/RDHAP

INTERVENTIONS:
Drug: Zanubrutinib and RCHOP/RDHAP — Alternating 3× R-CHOP/ 3× R-DHAOx, every 21 days plus oral Zanubrutinib in cycle 1, 3, 5 in combination with R-CHOP:
  R-CHOP (cycle 1,3,5):
  Rituximab 375 mg/m2 D1, I.V. Cyclophosphamide 750 mg/m2 D1, I.V. Doxorubicine 50 mg/m2 D1, I.V. Vincristine 1.4mg/m2(max 2mg)D1, I.V. Prednisone 100mg D1-5, oral Zanubrutinib 160mg BID D1-21, oral
  R-DHAP(cycle 2,4,6):
  Dexamethasone 40mg D1-4 oral/I.V. Rituximab 375mg/m2 D1, I.V. Ara-C 2×2g/m2 q12h D2, I.V. Cisplatin 100mg/m2 D1, I.V.
  Maintenance:
  Zanubrutinib, 160mg PO BID, rituximab 375mg/m2 repeated every 8 weeks, treatment will continue for up to 2 years or until progressive disease。

SUMMARY:
Evaluation the efficacy and safety of Zanubrutinib + R-CHOP/R-DHAP for the treatment mantle cell lymphoma.

DETAILED DESCRIPTION:
A single-arm, single-center, open-label phase II study of Zanubrutinib combined with R-CHOP/R-DHAP alternating induction therapy followed by Zanubrutinib rituximab maintenance therapy.The primary objective of this study was to assess CR and ORR rates after 6 cycles of initiation (i.e., at the end of induction therapy), and to collect adverse events during induction and maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of MCL according to WHO classification;
* Previously untreated MCL.
* Age ≥ 18 and ≤ 70 years old.
* ECOG, 0~2.
* Suitable for high-dose treatment including high-dose Ara-C.
* Stage II-IV (Ann Arbor).
* Measurable disease by computed tomography (CT)/magnetic resonance imaging (MRI). Measurable disease was defined as at least 1 lymph node > 1.5 cm in longest diameter and measurable in 2 perpendicular dimensions; in case of bone marrow infiltration only, bone marrow aspiration and biopsy are mandatory for all staging evaluations.
* The following laboratory tests during the screening period (unless related to MCL disease)
* 1) Neutrophils ≥1×109/L within 7 days prior to study entry, and no growth factor support therapy.
* 2) Platelets ≥75×109/L within 7 days prior to study entry without growth factor support or blood transfusion.
* 3) Hemoglobin ≥75g/L shall not be transfused within 7 days before the test. If bone marrow is involved, neutrophils ≥0.75×109/L, platelets ≥50×109/L, hemoglobin ≥50g/L)
* 4) Creatinine clearance ≥30ml/min
* 5) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3× upper limit of normal (ULN).
* International Standardized ratio (INR) ≤1.5 and activated partial prothrombin kinase time (APTT) ≤1.5×ULN. If there is a clotting factor inhibitor that causes an elevated INR or prolonged APTT, it is up to the investigator to decide whether to enroll the patient.
* Sexually active men and women of child-bearing potential must agree to use highly effective contraceptives (eg, condoms, implants, injectables, combined oral contraceptives, intrauterine devices, sexual abstinence, or sterilized partner) while on study; this should be maintained for 90 days after the last dose of study drug
* Life expectancy > 3 months.
* Written informed consent form according to GCP and national regulations.

Exclusion Criteria:

* Known CNS involvement of MCL, Leukemic non-lymphonodular mantle cell lymphoma was excluded.
* Major surgery within 4 weeks of screening
* Concomitant or previous malignancies within the last 2 years other than basal cell skin cancer or in situ uterine cervix cancer
* Clinically significant cardiovascular disease such as uncontrolled arrhythmias and hypertension , congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification or LVEF below 50%（AHA，2016）
* QTcF > 450 msec or other significant electrocardiogram (ECG) abnormalities including second-degree atrioventricular block Type II, or third-degree atrioventricular block
* Clinically significant hypersensitivity (eg, anaphylactic or anaphylactoid reactions to the compound of zanubrutinib itself or to the excipients in its formulation)
* Requires treatment with strong CYP3A inhibitors or strong CYP3A inducers
* Unable to swallow capsules or disease significantly affecting gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, bariatric surgery procedures, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction
* Active infection including infections requiring oral or intravenous antimicrobial therapy
* Patients with unresolved hepatitis B or C infection or known HIV positive infection
* History of stroke or intracranial hemorrhage within 6 months before first dose of study drug
* Pregnancy or lactation
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could have compromised the patient's safety, or put the study at risk
* Participation in another clinical trial within 30 days before enrollment in this study
* poor compliance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
CR rate after 6 cycles of induction therapy | 18 weeks
  To evaluate the CR rate after Zanubrutinib-based induction therapy in subjects with newly diagnosed MCL.

SECONDARY OUTCOMES:
ORR rate after 6 cycles of induction therapy | 18 weeks
  To evaluate the ORR rate after Zanubrutinib-based induction therapy in subjects with newly diagnosed MCL.
Progression free survival (PFS) | 60 weeks
  The time from start of treatment to progression or death from any cause
Overall survival (OS) | 60 weeks
  The time from start of treatment to death from any cause
duration of response, DOR | 60 weeks
  Defined as the time after the start of treatment from the first time remission criteria are met until disease progression or death is objectively recorded, whichever occurs first.
MRD negative rate at the end of induction therapy | 18 weeks
  MRD negative rate in peripheral blood or bone marrow at the end of induction therapy

CONTACTS AND LOCATIONS:
Overall Officials: Liping Su, M.D., Principal Investigator — Hematology Department of ShanXi Cancer Hospital
Locations (1):
- Hematology Department of ShanXi Cancer Hospital, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Plan to Share Clinical Study Report within six months after the study completed
Supporting Information: CSR
Time Frame: Within six months after the study completed
Access Criteria: Research site